CLINICAL TRIAL: NCT07273318
Title: Randomized, Open-Label, Comparative, Non-Profit Study to Evaluate the Performance and Safety of Osmonar® Medical Device Nasal Gel Versus Saline Solution in Patients With Dry Nose
Brief Title: Osmonar® Nasal Gel Versus Saline Solution in Patients With Dry Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Grasso (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor-Investigator, Michele Grasso, Principal Investigator, GIOVANNI PAOLO II Hospital of Lamezia Terme
Organization: GIOVANNI PAOLO II Hospital of Lamezia Terme (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMS/21/OSMONAR/01
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Dry Nose
Keywords: dry nose; medical device; randomized study; single-blind

STUDY DESIGN:
Intervention Model Description: randomized single-blind design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSMONAR Nasal Gel (Experimental): Medical Device Class IIa
  Interventions: Device: Osmonar
- Isotonic saline solution (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Osmonar — one application per nostril twice daily (in the morning and in the evening) administered for 14 consecutive days
  Arms: OSMONAR Nasal Gel
Other: Placebo — one application per nostril twice daily (in the morning and in the evening) administered for 14 consecutive days
  Arms: Isotonic saline solution

SUMMARY:
This study is being done to understand how well a medical device called OSMONAR Nasal Gel works and how safe it is for people who suffer from a dry nose.

A dry nose can cause discomfort, crusting, irritation, and breathing difficulties. There are not many effective treatments available. This study may help doctors find a new and safe option for people with this condition.

About 60 adults with symptoms of dry nose will take part.

* 30 people will use OSMONAR Nasal Gel
* 30 people will use a saline solution (a simple salt-water solution) Both groups will have similar symptoms. This helps doctors compare the two products fairly.

Each participant will use the assigned product for 14 days applying it twice a day as follows:

* once in each nostril in the morning
* once in each nostril in the evening

Each participant will have three visits:

* Visit 1 - Start of the study
* Visit 2 - Day 7
* Day 14 (End of treatment)

At each visit, the study doctor will:

* Perform a general medical check-up;
* Confirm the diagnosis of dry nose;
* Ask the participant to rate how dry their nose feels using a 10-cm Visual Analog Scale (VAS);
* Examine the inside of the nose using a fiber-optic rhinoscope to check for crusts, blockage, or breathing problems;
* Ask about satisfaction with the product and how easy it was to use;
* Check the participant's safety and whether the product is well tolerated.

The study will look at:

* How well symptoms improve.
* Changes in nasal dryness and discomfort.
* How the inside of the nose looks during examination.
* How safe and well tolerated the treatment is.
* How satisfied participants are with the treatment.

This study was planned, organized, and performed autonomously as a non-profit study without any external support by the principal investigator of the Otorhinolaryngology Department at Giovanni Paolo II Hospital in Lamezia Terme.

The results of the study will help doctors learn whether OSMONAR Nasal Gel can be a safe and effective treatment for people with dry nose and whether it works better than saline solution:

DETAILED DESCRIPTION:
Nasal dryness is a frequent condition caused by mucosal atrophy, chronic irritation, infections, environmental factors, or systemic diseases such as Sjögren's syndrome. Symptoms may include crusting, nasal obstruction, irritation, and breathing discomfort. Management typically involves eliminating triggering factors, maintaining hydration, humidifying the environment, and using topical agents such as saline solutions, oils, or hyaluronic-acid-based products.

This study evaluates the performance and safety of OSMONAR Nasal Gel, a medical device containing pyrohyaluronate (PCA) and hyaluronic acid (HA). The product is designed to hydrate the nasal mucosa, form a protective film against external irritants, and support mucosal repair. The aim is to determine whether OSMONAR can improve symptoms associated with dry nose more effectively than saline solution.

A total of 60 adults with dry nose syndrome will be randomized into two groups:

* OSMONAR Nasal Gel: one application per nostril twice daily for 14 days;
* Placebo (Isotonic saline solution): 1 application per nostril twice daily for 14 days.

The study is randomized and single-blind and includes three visits: baseline (Day 0), interim (Day 7), and final evaluation (Day 14). At each visit, participants will rate nasal dryness using a 10-cm Visual Analog Scale (VAS). In addition, nasal crusting, obstruction, and respiratory discomfort will be assessed by Investigator using fiber-optic rhinoscopy. Safety will be evaluated by monitoring adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Patients affected by dry nose;
3. Willing to comply with study requirements, using the tested products for 14 consecutive days;
4. Readiness not to participate in another clinical study during this study;
5. Commitment to using contraceptive methods (for women of childbearing age only);
6. Negative pregnancy testing (beta human chorionic gonadotropin test in urine) at baseline (only for women in childbearing age);
7. Written informed consent by the participant.

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the OSMONAR or of saline solution; 4. Lesions/infections in the nasal area;

5. Use of preparations that may influence the study outcome within the last 2 weeks prior to baseline and during the study (e.g. antibiotics, corticosteroids etc.);

6. History or presence of any other clinically significant known (self-reported) condition /disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject;

7. Pregnancy, nursing or within first 3 months post-partum;

8. History of or current abuse of drugs, alcohol or medication;

9. Participation in another study during the last 30 days prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Subjective nasal dryness | 14 days
  The change in subjective nasal dryness, as evaluated by the patient using a Visual Analogue Scale (VAS) score ranging from 0 (no nasal dryness) to 10 (maximum level of nasal dryness), will be assessed from baseline to final visit (day 14). The mean values will be compared between the two treatment groups
Incidence of adverse events | 14 days
  The incidence of adverse events (AEs), serious adverse events (SAEs), adverse device effects (ADEs), and serious adverse device effects (SADEs) will be collected by Investigators, compared between the two groups, and analyzed with the incidence in standard population

SECONDARY OUTCOMES:
Presence of nasal crusts | 14 days
  Percentage of subjects with nasal crusts evaluated by fiber-optic rhinoscopy at baseline and at Final Visit (day 14). The decrease in % will be compared between the two treatment groups
Presence of nasal obstruction | 14 days
  Percentage of subjects with nasal obstruction evaluated by fiber-optic rhinoscopy at baseline and at Final Visit (day 14). The decrease in % will be compared between the two treatment groups
Presence of respiratory discomfort | 14 days
  Percentage of subjects with respiratory discomfort evaluated by fiber-optic rhinoscopy at baseline and at Final Visit (day 14). The decrease in % will be compared between the two treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Michele Grasso, Dr., Principal Investigator — Presidio Ospedaliero di Lamezia Terme Giovanni Paolo II
Locations (1):
- Department of Otolaryngology - Presidio Ospedaliero di Lamezia Terme Giovanni Paolo II, Lamezia Terme, CZ, Italy

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) that underlie results in a publication
Supporting Information: CSR
Time Frame: IPD will be available from the corresponding author, upon reasonable request after the result publication.
Access Criteria: Other researchers will receive the IPD upon reasonable request from the corresponding author.